CLINICAL TRIAL: NCT04699994
Title: Multicenter Phase II Trial to Evaluate the Safety and Efficacy of FLOT Therapy for Resectable Esophageal Squamous Cell Carcinoma (Preoperative FLOT PII)
Brief Title: Prospective Trial to Evaluate the Safety and Efficacy to Treat Esophageal Cancer Using 5-FU, Oxaliplatin, and Docetaxel
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Keio University (Other)
Responsible Party: Principal Investigator, Hirofumi Kawakubo, Associate Professor, Keio University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N20190007
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FLOT therapy (Experimental)
  Interventions: Drug: FLOT therapy

INTERVENTIONS:
Drug: FLOT therapy — Preoperative FLOT therapy

SUMMARY:
The current multicenter prospective phase II study aims to evaluate the safety and efficacy of preoperative FLOT therapy for esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically diagnosed as esophageal squamous cell carcinoma (squamous, adenosquamous, basaloid)
2. Primary tumor is located mainly in the thoracic esophagus
3. cT1N1-3M0-1 (only supraclavicular LN metastasis is included as M1), cT2-3N0-3M0-1 (only supraclavicular LN metastasis is included as M1)
4. Twenty years old or older as of registration
5. Performance status (PS) 0 or 1
6. Patients have target lesions
7. No previous history of esophageal cancer except for the followings

1) pT1a-LPM (M2) or deeper following EMR/ESD 2) pT1a-MM (M3) with vascular invasion following EMR/ ESD 8. No previous history of chemotherapy/radiotherapy/endocrine therapy except for hormone therapy for prostate cancer after 5 years interval 9. Patients who meet the following criteria

1. Neutrophil > 1,500 /mm3
2. Platelet > 10.0x10^4 /mm3
3. Hb ≧9.0 g/dL
4. Total bilirubin ≦ 1.5 mg/dL
5. AST ≦ 100 IU/L
6. ALT ≦ 100 IU/L
7. SpO2 ≧ 95 %
8. Creatinine clearance ≧ 50 mL/min 10. Patients who can undergo esophagectomy 11. Agree with the participation to the current study

Exclusion Criteria:

1. Patients who received any treatment for cancer within 3 years
2. Patients who have active infectious diseases
3. HBs Ag positive or HIV Ab positive
4. Pregnant or breast feeding
5. Patients with psychological disorder
6. On systemic steroid therapy
7. Require flucytocine, phenytoin, warfarin
8. Allergic to iodine
9. Allergic to DTX, LOHP, polisorbate 80
10. Uncontrollable diabetes
11. Severe COPD or lung fibrosis
12. Severe hypertension
13. Unstable angina
14. Patients whom investigators evaluate as ineligible

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-25 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Histological response rate (Grade 2 or 3 in Japanese Classification of Esophageal Cancer, 11th Edition) | 2.5 years

SECONDARY OUTCOMES:
Response rate | 2.5 years
Histological complete response rate | 2.5 years
Treatment completion rate | 2.5 years
Curative resection rate | 2.5 years
Recurrence free survival | 4.5 years
Overall survival | 4.5 years
Incidence rate of adverse event during FLOT | 2.5 years
Perioperative complication rate | 2.5 years
Late phase complication rate | 4.5 years
Incidence rate of severe adverse event | 2.5 years
Incidence rate of all adverse event | 4.5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Keio University Hospital, Tokyo, Japan